CLINICAL TRIAL: NCT04267133
Title: Home-based Videoplethysmographic Detection of Atrial Fibrillation
Brief Title: Video-based Detection of Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Jean-Philippe Couderc, Associate Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 68409
Record Dates: First submitted 2020-02-10; First posted 2020-02-12 (Actual); Results first posted 2023-01-27 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- All Participants (Experimental)
  Interventions: Diagnostic Test: Facial video of detection of cardiac disease

INTERVENTIONS:
Diagnostic Test: Facial video of detection of cardiac disease — This project proposes to evaluate a non-contact video recording technology to detect the presence of AF. The technology extracts a pulsatile signal by measuring the subtle variations in skin color of a patient's face (flushing) due to the variations of blood volume underneath the skin. The technology uses a standard web camera. This technique is videoplethysmography (VPG).

SUMMARY:
The project focuses on the evaluation of a novel, contactless monitoring technology to measure the blood pulsatile signal based on the video recording of an individual's face. The variability of the pulse rate is computed to identify the presence of atrial fibrillation (AF). We propose to enroll 315 patients with symptomatic AF, paroxysmal or persistent, who go through successful radiofrequency ablation or electrical cardioversion. A computer tablet will be used by the subjects at home during 14 days after their procedure to read emails, browse the internet and watch videos. Facial video recordings will be automatically acquired during these daily activities by the tablet device. The subject will be wearing an ECG patch during the follow-up period. The one-lead continuous ECG will be used as a reference to verify the presence of AF rhythm during facial video recordings. The primary aim of the study is to demonstrate the validity and robustness of the video-based technology to detect the presence of AF when facial videos are acquired by the patients at home.

ELIGIBILITY:
Inclusion Criteria:

* Men and women older than 18 years of age,
* Medically-managed for symptomatic AF (persistent or paroxysmal),
* In sinus rhythm after their ablation procedure,
* In sinus rhythm after trans-thoracic electrical cardioversion.

Exclusion Criteria:

* Implanted with a device (pacemaker, CRT, ICD) and a ventricular pacing requirement superior or equal to 70%,
* Known allergic reaction to adhesives or hydrogels or with a family history of adhesive skin allergies,
* Unable to cooperate with the protocol due to dementia, psychological, or other related reason,
* Refusing to sign the consent for participation,
* Unable to operate the device such as blind patients.
* Patients with Parkinson disease (or other central nervous system disorder/Tremor) who cannot record a stable video signal of their face.
* The subject was previously enrolled in the current study.
* The subject wears clothing covering the face, or uses facial makeup that will interfere with the quality of facial recordings.
* Subject does not have internet access at home and lacks the technology to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2018-05-24 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Strong Memorial Hospital, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benjamin EJ, Chen PS, Bild DE, Mascette AM, Albert CM, Alonso A, Calkins H, Connolly SJ, Curtis AB, Darbar D, Ellinor PT, Go AS, Goldschlager NF, Heckbert SR, Jalife J, Kerr CR, Levy D, Lloyd-Jones DM, Massie BM, Nattel S, Olgin JE, Packer DL, Po SS, Tsang TS, Van Wagoner DR, Waldo AL, Wyse DG. Prevention of atrial fibrillation: report from a national heart, lung, and blood institute workshop. Circulation. 2009 Feb 3;119(4):606-18. doi: 10.1161/CIRCULATIONAHA.108.825380. PMID 19188521
- [Background] Jabaudon D, Sztajzel J, Sievert K, Landis T, Sztajzel R. Usefulness of ambulatory 7-day ECG monitoring for the detection of atrial fibrillation and flutter after acute stroke and transient ischemic attack. Stroke. 2004 Jul;35(7):1647-51. doi: 10.1161/01.STR.0000131269.69502.d9. Epub 2004 May 20. PMID 15155965
- [Background] Tayal AH, Tian M, Kelly KM, Jones SC, Wright DG, Singh D, Jarouse J, Brillman J, Murali S, Gupta R. Atrial fibrillation detected by mobile cardiac outpatient telemetry in cryptogenic TIA or stroke. Neurology. 2008 Nov 18;71(21):1696-701. doi: 10.1212/01.wnl.0000325059.86313.31. Epub 2008 Sep 24. PMID 18815386
- [Background] Healey JS, Connolly SJ, Gold MR, Israel CW, Van Gelder IC, Capucci A, Lau CP, Fain E, Yang S, Bailleul C, Morillo CA, Carlson M, Themeles E, Kaufman ES, Hohnloser SH; ASSERT Investigators. Subclinical atrial fibrillation and the risk of stroke. N Engl J Med. 2012 Jan 12;366(2):120-9. doi: 10.1056/NEJMoa1105575. PMID 22236222
- [Background] Sanna T, Diener HC, Passman RS, Di Lazzaro V, Bernstein RA, Morillo CA, Rymer MM, Thijs V, Rogers T, Beckers F, Lindborg K, Brachmann J; CRYSTAL AF Investigators. Cryptogenic stroke and underlying atrial fibrillation. N Engl J Med. 2014 Jun 26;370(26):2478-86. doi: 10.1056/NEJMoa1313600. PMID 24963567
- [Background] Verkruysse W, Svaasand LO, Nelson JS. Remote plethysmographic imaging using ambient light. Opt Express. 2008 Dec 22;16(26):21434-45. doi: 10.1364/oe.16.021434. PMID 19104573
- [Background] Couderc JP, Kyal S, Mestha LK, Xu B, Peterson DR, Xia X, Hall B. Detection of atrial fibrillation using contactless facial video monitoring. Heart Rhythm. 2015 Jan;12(1):195-201. doi: 10.1016/j.hrthm.2014.08.035. Epub 2014 Aug 29. PMID 25179488
- [Background] Oral H, Knight BP, Ozaydin M, Tada H, Chugh A, Hassan S, Scharf C, Lai SW, Greenstein R, Pelosi F Jr, Strickberger SA, Morady F. Clinical significance of early recurrences of atrial fibrillation after pulmonary vein isolation. J Am Coll Cardiol. 2002 Jul 3;40(1):100-4. doi: 10.1016/s0735-1097(02)01939-3. PMID 12103262
- [Background] Lee SH, Tai CT, Hsieh MH, Tsai CF, Lin YK, Tsao HM, Yu WC, Huang JL, Ueng KC, Cheng JJ, Ding YA, Chen SA. Predictors of early and late recurrence of atrial fibrillation after catheter ablation of paroxysmal atrial fibrillation. J Interv Card Electrophysiol. 2004 Jun;10(3):221-6. doi: 10.1023/B:JICE.0000026915.02503.92. PMID 15133358
- [Background] Chang SL, Tsao HM, Lin YJ, Lo LW, Hu YF, Tuan TC, Suenari K, Tai CT, Li CH, Chao TF, Lin YK, Tsai CF, Wu TJ, Chen SA. Characteristics and significance of very early recurrence of atrial fibrillation after catheter ablation. J Cardiovasc Electrophysiol. 2011 Nov;22(11):1193-8. doi: 10.1111/j.1540-8167.2011.02095.x. Epub 2011 May 26. PMID 21615812
- [Background] Andrade JG, Khairy P, Verma A, Guerra PG, Dubuc M, Rivard L, Deyell MW, Mondesert B, Thibault B, Talajic M, Roy D, Macle L. Early recurrence of atrial tachyarrhythmias following radiofrequency catheter ablation of atrial fibrillation. Pacing Clin Electrophysiol. 2012 Jan;35(1):106-16. doi: 10.1111/j.1540-8159.2011.03256.x. Epub 2011 Nov 6. PMID 22054110
- [Background] Bianconi L, Mennuni M, Lukic V, Castro A, Chieffi M, Santini M. Effects of oral propafenone administration before electrical cardioversion of chronic atrial fibrillation: a placebo-controlled study. J Am Coll Cardiol. 1996 Sep;28(3):700-6. doi: 10.1016/0735-1097(96)00230-6. PMID 8772759
- [Background] Siaplaouras S, Jung J, Buob A, Heisel A. Incidence and management of early recurrent atrial fibrillation (ERAF) after transthoracic electrical cardioversion. Europace. 2004 Jan;6(1):15-20. doi: 10.1016/j.eupc.2003.09.010. PMID 14697721
- [Background] Yu WC, Lin YK, Tai CT, Tsai CF, Hsieh MH, Chen CC, Hsu TL, Ding YA, Chang MS, Chen SA. Early recurrence of atrial fibrillation after external cardioversion. Pacing Clin Electrophysiol. 1999 Nov;22(11):1614-9. doi: 10.1111/j.1540-8159.1999.tb00380.x. PMID 10598964
- [Background] Moller M, Torp-Pedersen CT, Kober L. Dofetilide in patients with congestive heart failure and left ventricular dysfunction: safety aspects and effect on atrial fibrillation. The Danish Investigators of Arrhythmia and Mortality on Dofetilide (DIAMOND) Study Group. Congest Heart Fail. 2001 May-Jun;7(3):146-150. doi: 10.1111/j.1527-5299.2001.00243.x. PMID 11828153
- [Background] Turakhia MP, Ullal AJ, Hoang DD, Than CT, Miller JD, Friday KJ, Perez MV, Freeman JV, Wang PJ, Heidenreich PA. Feasibility of extended ambulatory electrocardiogram monitoring to identify silent atrial fibrillation in high-risk patients: the Screening Study for Undiagnosed Atrial Fibrillation (STUDY-AF). Clin Cardiol. 2015 May;38(5):285-92. doi: 10.1002/clc.22387. Epub 2015 Apr 14. PMID 25873476
- [Background] Tung CE, Su D, Turakhia MP, Lansberg MG. Diagnostic Yield of Extended Cardiac Patch Monitoring in Patients with Stroke or TIA. Front Neurol. 2015 Jan 12;5:266. doi: 10.3389/fneur.2014.00266. eCollection 2014. PMID 25628595
- [Background] Rosenberg MA, Samuel M, Thosani A, Zimetbaum PJ. Use of a noninvasive continuous monitoring device in the management of atrial fibrillation: a pilot study. Pacing Clin Electrophysiol. 2013 Mar;36(3):328-33. doi: 10.1111/pace.12053. Epub 2012 Dec 13. PMID 23240827
- [Background] Chen LY, Agarwal SK, Norby FL, Gottesman RF, Loehr LR, Soliman EZ, Mosley TH, Folsom AR, Coresh J, Alonso A. Persistent but not Paroxysmal Atrial Fibrillation Is Independently Associated With Lower Cognitive Function: ARIC Study. J Am Coll Cardiol. 2016 Mar 22;67(11):1379-80. doi: 10.1016/j.jacc.2015.11.064. No abstract available. PMID 26988962
- [Background] Couderc JP. The Telemetric and Holter ECG Warehouse (THEW): the first three years of development and research. J Electrocardiol. 2012 Nov-Dec;45(6):677-83. doi: 10.1016/j.jelectrocard.2012.08.001. Epub 2012 Sep 28. PMID 23022305
- [Background] Couderc JP. The telemetric and Holter ECG warehouse initiative (THEW): a data repository for the design, implementation and validation of ECG-related technologies. Annu Int Conf IEEE Eng Med Biol Soc. 2010;2010:6252-5. doi: 10.1109/IEMBS.2010.5628067. PMID 21097349
- [Derived] Dzikowicz DJ, Aktas M, Mykins B, Xia X, Zareba W, Couderc JP. Identifying Demographic Factors Affecting the ECG Duration Collected Using a Single-Lead ECG Patch Device. Ann Noninvasive Electrocardiol. 2025 May;30(3):e70068. doi: 10.1111/anec.70068. PMID 40320720

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Participants
Started | 256
Completed | 251
Not Completed | 5
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 4

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 255
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85
  Male | 170
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 245
  Unknown or Not Reported | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 249
  More than one race | 2
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 255

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Receiver Operating Characteristic Curve (AUC) for the Detection of Atrial Fibrillation
Description: The outcome measure is the AUC of the curve obtained from the ROC analysis. The curve is a combination of specificity and sensitivity of detecting atrial fibrillation. The range of the curve is 0.5-1.0 where 0.5 would be random detection of atrial fibrillation and 1.0 would be perfect performance.
Time Frame: 2 weeks
Population: We collected data for the AUC from 108 patients. We collected 977 recordings from these 108 patients.
Measure: Number; unit: probability
Arm/Group | All Participants
Number analyzed (Participants) | 108
probability | 0.74

ADVERSE EVENTS:
Time Frame: 15 days
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/256
Serious Adverse Events (participants affected / at risk) | 0/256
Other Adverse Events (participants affected / at risk) | 0/256

LIMITATIONS AND CAVEATS:
We did not fully enroll the sample size needed to reach statistical significance.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-07-02): https://cdn.clinicaltrials.gov/large-docs/33/NCT04267133/Prot_SAP_000.pdf
  • Informed Consent Form (2020-06-03): https://cdn.clinicaltrials.gov/large-docs/33/NCT04267133/ICF_001.pdf